CLINICAL TRIAL: NCT05250778
Title: Room Design Nudge on Hospitalist Bedside Etiquette and Patient Satisfaction
Brief Title: Nudges on Hospitalist Behavior and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Sumarsono, Assistant Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STU-2021-1057
Record Dates: First submitted 2022-02-01; First posted 2022-02-22 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Patient Satisfaction; Etiquette, Medical
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nudge Group (Experimental): Encounters in this group will be nudged
  Interventions: Behavioral: Nudge
- Control Group (No Intervention): Encounters in this group will not receive a nudge.

INTERVENTIONS:
Behavioral: Nudge — Room intervention
  Arms: Nudge Group

SUMMARY:
Physician behavior plays an important role on patient perception of their care team and on patient satisfaction. Though studies have attempted to impact how physicians interact with their patients through various initiatives, the effect of more subtle nudges on physician behavior have not been studies. As such, the investigators propose a randomized controlled deception trial to evaluate the impact of nudges on hospitalist behavior and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalist Physicians at Parkland Memorial Hospital who are willing to participate

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Physician Sitting Rate | During the Observed Physician Encounter
  This will be a binary measurement of whether or not the physician sits with the patient during the observed encounter.

SECONDARY OUTCOMES:
TAISCH: Tool to Assess Inpatient Satisfaction with Care from Hospitalists | Immediately Following Observed Physician Encounter
  This is a previously validated measure of patient satisfaction for hospitalists.

CONTACTS AND LOCATIONS:
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iyer R, Park D, Kim J, Newman C, Young A, Sumarsono A. Effect of chair placement on physicians' behavior and patients' satisfaction: randomized deception trial. BMJ. 2023 Dec 15;383:e076309. doi: 10.1136/bmj-2023-076309. PMID 38101923